CLINICAL TRIAL: NCT01817127
Title: Functional Deconstruction of Human Milk Oligosaccharides and Lipids
Brief Title: Elucidation of Breast Milk Composition and Structure Over the First Year of Lactation: UC Davis Lactation Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: California Dairy Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 216198
Record Dates: First submitted 2013-03-11; First posted 2013-03-22 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Gestational Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast milk, blood, saliva, urine, stool, epidermal skin cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Main Study: Women enrolled in this cohort of the study will collect their breast milk, infant urine and stool, and their urine and stool samples. Blood and saliva will be collected from these participants by study personnel.
- Gestational Diabetes Mellitus Cohort: Women who have been diagnosed with gestational diabetes mellitus, type 2 diabetes mellitus or impaired glucose tolerance will be enrolled in this cohort. Participants will be asked to report their fasting and postprandial blood glucose levels if they are monitoring these outcomes at home with a glucometer.
- Fresh Milk Cohort: Women enrolled in this cohort will provide fresh milk samples (stored in the refrigerator and picked up by study personnel within 1 hour of collection) for analysis of glycan composition and gene expression of glycan metabolizing enzymes of somatic cells in milk.
- RNA Milk Fat Cohort: Women enrolled in this cohort must have given birth to sons and will collect a fresh milk sample for transcriptomic analysis compared against non-human primate milk.
- Skin Study: This cohort includes mothers and their infants who will provide milk and infant stratum corneum cells to act as the control group for a different study designed to investigate skin function in premature infants.
- BMMI Project: Subjects enrolled in this cohort will be part of the control group for the BMMI Project.

SUMMARY:
This observational study is designed to determine how sugars, lipids and proteins in breast milk vary among mothers; is affected by maternal diet, health and microbiota and vary over the course of lactation. Additionally, the study is designed to determine how the structure and composition of complex milk sugars, maternal health status and diet influence the development and maintenance of infant gut microflora.

DETAILED DESCRIPTION:
This study's objectives include: 1) develop a better understanding of the composition and structures of breast milk over the early stages of lactation with specific emphasis on the glycans and lipids; 2) how glycan diversity relates to maternal and infant gut microbiota with an emphasis on bifidobacteria species; 3)how milk composition and structure relate to maternal health and diet.

These samples will be analyzed using comprehensive gas and liquid chromatographic methods, nuclear magnetic resonance (NMR) spectroscopy and mass spectrometry (MS); and next generation sequencing, terminal restriction fragment length polymorphism and quantitative polymerase chain reaction.

There are several cohorts to the main study.

Gestational Diabetes Mellitus Cohort. The aim of this study is to investigate the differences between milk composition, infant and maternal gut microbiota from women with and without gestational diabetes mellitus or type 2 diabetes vs. controls.

Fresh Milk Study. The aim of this study is to elucidate the relationship between the expression of glycan metabolizing genes of mammary epithelial cells and levels of milk glycans.

RNA Study. The aim of this study is to compare the RNA of milk fat globule membrane crescents in human milk against epithelial expression profiles in non-human primate milk.

Skin Study. The aim of this study is to provide skin samples from healthy term infants to act as the control group for a different study with preterm infants.

Breast Milk, Gut Microbiome, and Immunity (BMMI) Project. The aim of this study is to provide healthy control samples for the BMMI project. The BMMI project is a multi-investigative project designed to elucidate how maternal nutrient status, and milk composition and structure influence infant gut microbiome from participants in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years and older who plan to breastfeed for at least 6 months
* Women who are in good health
* Women with or without diagnosis of gestational diabetes mellitus, or type 2 diabetes mellitus or impaired glucose tolerance

Exclusion Criteria:

* Women who do not plan to breastfeed for at least 6 months
* Women who give birth to pre-term infants
* Women who smoke, either currently or 1 year before becoming pregnant
* Women who have chronic medical conditions or communicable diseases
* Women who take metabolic altering drugs such as corticosteroids or thyroid medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women and women diagnosed with gestational diabetes mellitus or type 2 diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2028-09-04 (Estimated)

PRIMARY OUTCOMES:
Human milk glycans | Change from day 2 to day 366
  Human milk glycans: human milk oligosaccharides and glycoconjugates to lipids, proteins and peptides will be measured by MS methods.

SECONDARY OUTCOMES:
Microbiota | 3rd trimester pregnancy and Day 2-Day 366 postpartum
  Maternal and infant gut microbiota, infant skin microbiota will be measured using next generation sequencing, terminal restriction fragment length polymorphism and quantitative polymerase chain reaction.
Proteome | Day 2-Day 366 postpartum
  Milk and infant stratum corneum will be analyzed by MS methods.
Lipidome | Day 2-Day 366 postpartum
  Milk and skin will be analyzed by gas chromatography and MS methods.
Maternal plasma lipids | 3rd trimester pregnancy and 2 months postpartum
  The plasma lipid profile will be analyzed by enzyme assay by UC Davis Pathology Lab.
Peptidome | 3rd trimester pregnancy and Day 2-Day 366
  Milk and infant and maternal stool will be analyzed by MS methods.
Metabolome by Nuclear Magnetic Spectroscopy (NMR) | 3rd trimester of pregnancy and D2-Day 366
  Milk, maternal and infant urine and stool will be analyzed by NMR spectroscopy.
Metabolome by MS | Day 2-Day 366 postpartum
  Milk, maternal and infant urine and stool will be analyzed by MS.
Secretor status genotyping | 3rd trimester pregnancy and Day 60 postpartum
  Maternal secretor status genotyping will be determined by quantitative polymerase chain reaction for the functional fucosyltransferase 2 gene from maternal saliva.
Maternal fasting and postprandial blood sugar | 3rd trimester of pregnancy and Day 3-7
  Maternal blood sugar will be checked by finger stick using a glucometer in women diagnosed with gestational diabetes mellitus.
Maternal plasma lipoprotein size distribution | 3rd trimester of pregnancy and Day 60 postpartum
  Plasma lipoprotein size distribution and concentration will be analyzed by NMR spectroscopy by LipoScience.
Human Milk Transcriptomics | 3 and 6 months postpartum
  Milk samples will be preserved with RNA-later, RNA extracted and analyzed by next generation sequencing techniques.

OTHER OUTCOMES:
Alkaline phosphatase levels | Days 2 through 50
  Milk samples will be analyzed for alkaline phosphatase activity by fluorometric assay

CONTACTS AND LOCATIONS:
Overall Officials: Bruce German, PhD, Principal Investigator — University of California, Davis; Carlito Lebrilla, PhD, Principal Investigator — University of California, Davis; David Mills, PhD, Principal Investigator — University of California, Davis; Bart Weimer, PhD, Principal Investigator — University of California, Davis; Xiangdong Wu, PhD, Principal Investigator — University of California, Davis; Helen Raybould, PhD, Principal Investigator — University of California, Davis; Jennifer T. Smilowitz, PhD, Principal Investigator — University of California, Davis; Danielle Lemay, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

REFERENCES:
- [Background] Totten SM, Zivkovic AM, Wu S, Ngyuen U, Freeman SL, Ruhaak LR, Darboe MK, German JB, Prentice AM, Lebrilla CB. Comprehensive profiles of human milk oligosaccharides yield highly sensitive and specific markers for determining secretor status in lactating mothers. J Proteome Res. 2012 Dec 7;11(12):6124-33. doi: 10.1021/pr300769g. Epub 2012 Nov 19. PMID 23140396
- [Background] De Leoz ML, Gaerlan SC, Strum JS, Dimapasoc LM, Mirmiran M, Tancredi DJ, Smilowitz JT, Kalanetra KM, Mills DA, German JB, Lebrilla CB, Underwood MA. Lacto-N-tetraose, fucosylation, and secretor status are highly variable in human milk oligosaccharides from women delivering preterm. J Proteome Res. 2012 Sep 7;11(9):4662-72. doi: 10.1021/pr3004979. Epub 2012 Aug 28. PMID 22900748
- [Background] Neville MC, Anderson SM, McManaman JL, Badger TM, Bunik M, Contractor N, Crume T, Dabelea D, Donovan SM, Forman N, Frank DN, Friedman JE, German JB, Goldman A, Hadsell D, Hambidge M, Hinde K, Horseman ND, Hovey RC, Janoff E, Krebs NF, Lebrilla CB, Lemay DG, MacLean PS, Meier P, Morrow AL, Neu J, Nommsen-Rivers LA, Raiten DJ, Rijnkels M, Seewaldt V, Shur BD, VanHouten J, Williamson P. Lactation and neonatal nutrition: defining and refining the critical questions. J Mammary Gland Biol Neoplasia. 2012 Jun;17(2):167-88. doi: 10.1007/s10911-012-9261-5. Epub 2012 Jul 1. PMID 22752723
- [Background] Garrido D, Nwosu C, Ruiz-Moyano S, Aldredge D, German JB, Lebrilla CB, Mills DA. Endo-beta-N-acetylglucosaminidases from infant gut-associated bifidobacteria release complex N-glycans from human milk glycoproteins. Mol Cell Proteomics. 2012 Sep;11(9):775-85. doi: 10.1074/mcp.M112.018119. Epub 2012 Jun 27. PMID 22745059
- [Background] Sela DA, Garrido D, Lerno L, Wu S, Tan K, Eom HJ, Joachimiak A, Lebrilla CB, Mills DA. Bifidobacterium longum subsp. infantis ATCC 15697 alpha-fucosidases are active on fucosylated human milk oligosaccharides. Appl Environ Microbiol. 2012 Feb;78(3):795-803. doi: 10.1128/AEM.06762-11. Epub 2011 Dec 2. PMID 22138995
- [Background] Marcobal A, Barboza M, Sonnenburg ED, Pudlo N, Martens EC, Desai P, Lebrilla CB, Weimer BC, Mills DA, German JB, Sonnenburg JL. Bacteroides in the infant gut consume milk oligosaccharides via mucus-utilization pathways. Cell Host Microbe. 2011 Nov 17;10(5):507-14. doi: 10.1016/j.chom.2011.10.007. Epub 2011 Oct 27. PMID 22036470
- [Background] Froehlich JW, Barboza M, Chu C, Lerno LA Jr, Clowers BH, Zivkovic AM, German JB, Lebrilla CB. Nano-LC-MS/MS of glycopeptides produced by nonspecific proteolysis enables rapid and extensive site-specific glycosylation determination. Anal Chem. 2011 Jul 15;83(14):5541-7. doi: 10.1021/ac2003888. Epub 2011 Jun 28. PMID 21661761
- [Background] Sela DA, Li Y, Lerno L, Wu S, Marcobal AM, German JB, Chen X, Lebrilla CB, Mills DA. An infant-associated bacterial commensal utilizes breast milk sialyloligosaccharides. J Biol Chem. 2011 Apr 8;286(14):11909-18. doi: 10.1074/jbc.M110.193359. Epub 2011 Feb 2. PMID 21288901
- [Background] Nwosu CC, Strum JS, An HJ, Lebrilla CB. Enhanced detection and identification of glycopeptides in negative ion mode mass spectrometry. Anal Chem. 2010 Dec 1;82(23):9654-62. doi: 10.1021/ac101856r. Epub 2010 Nov 4. PMID 21049935
- [Background] Zivkovic AM, German JB, Lebrilla CB, Mills DA. Human milk glycobiome and its impact on the infant gastrointestinal microbiota. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4653-8. doi: 10.1073/pnas.1000083107. Epub 2010 Aug 2. PMID 20679197
- [Background] Froehlich JW, Dodds ED, Barboza M, McJimpsey EL, Seipert RR, Francis J, An HJ, Freeman S, German JB, Lebrilla CB. Glycoprotein expression in human milk during lactation. J Agric Food Chem. 2010 May 26;58(10):6440-8. doi: 10.1021/jf100112x. PMID 20415418
- [Background] Marcobal A, Barboza M, Froehlich JW, Block DE, German JB, Lebrilla CB, Mills DA. Consumption of human milk oligosaccharides by gut-related microbes. J Agric Food Chem. 2010 May 12;58(9):5334-40. doi: 10.1021/jf9044205. PMID 20394371
- [Background] Ninonuevo MR, Ward RE, LoCascio RG, German JB, Freeman SL, Barboza M, Mills DA, Lebrilla CB. Methods for the quantitation of human milk oligosaccharides in bacterial fermentation by mass spectrometry. Anal Biochem. 2007 Feb 1;361(1):15-23. doi: 10.1016/j.ab.2006.11.010. Epub 2006 Nov 27. PMID 17181994
- [Background] Locascio RG, Ninonuevo MR, Kronewitter SR, Freeman SL, German JB, Lebrilla CB, Mills DA. A versatile and scalable strategy for glycoprofiling bifidobacterial consumption of human milk oligosaccharides. Microb Biotechnol. 2009 May;2(3):333-42. doi: 10.1111/j.1751-7915.2008.00072.x. Epub 2008 Dec 5. PMID 21261928
- [Background] Ninonuevo MR, Perkins PD, Francis J, Lamotte LM, LoCascio RG, Freeman SL, Mills DA, German JB, Grimm R, Lebrilla CB. Daily variations in oligosaccharides of human milk determined by microfluidic chips and mass spectrometry. J Agric Food Chem. 2008 Jan 23;56(2):618-26. doi: 10.1021/jf071972u. Epub 2007 Dec 19. PMID 18088092
- [Background] LoCascio RG, Ninonuevo MR, Freeman SL, Sela DA, Grimm R, Lebrilla CB, Mills DA, German JB. Glycoprofiling of bifidobacterial consumption of human milk oligosaccharides demonstrates strain specific, preferential consumption of small chain glycans secreted in early human lactation. J Agric Food Chem. 2007 Oct 31;55(22):8914-9. doi: 10.1021/jf0710480. Epub 2007 Oct 5. PMID 17915960
- [Background] Ninonuevo MR, Park Y, Yin H, Zhang J, Ward RE, Clowers BH, German JB, Freeman SL, Killeen K, Grimm R, Lebrilla CB. A strategy for annotating the human milk glycome. J Agric Food Chem. 2006 Oct 4;54(20):7471-80. doi: 10.1021/jf0615810. PMID 17002410
- [Background] Chu CS, Ninonuevo MR, Clowers BH, Perkins PD, An HJ, Yin H, Killeen K, Miyamoto S, Grimm R, Lebrilla CB. Profile of native N-linked glycan structures from human serum using high performance liquid chromatography on a microfluidic chip and time-of-flight mass spectrometry. Proteomics. 2009 Apr;9(7):1939-51. doi: 10.1002/pmic.200800249. PMID 19288519
- [Background] Hong P, Ninonuevo MR, Lee B, Lebrilla C, Bode L. Human milk oligosaccharides reduce HIV-1-gp120 binding to dendritic cell-specific ICAM3-grabbing non-integrin (DC-SIGN). Br J Nutr. 2009 Feb;101(4):482-6. doi: 10.1017/s0007114508025804. PMID 19230080
- [Background] Lewis ZT, Bokulich NA, Kalanetra KM, Ruiz-Moyano S, Underwood MA, Mills DA. Use of bifidobacterial specific terminal restriction fragment length polymorphisms to complement next generation sequence profiling of infant gut communities. Anaerobe. 2013 Feb;19:62-9. doi: 10.1016/j.anaerobe.2012.12.005. Epub 2012 Dec 20. PMID 23261904
- [Background] Garrido D, Ruiz-Moyano S, Jimenez-Espinoza R, Eom HJ, Block DE, Mills DA. Utilization of galactooligosaccharides by Bifidobacterium longum subsp. infantis isolates. Food Microbiol. 2013 Apr;33(2):262-70. doi: 10.1016/j.fm.2012.10.003. Epub 2012 Oct 22. PMID 23200660
- [Background] Gordon JI, Dewey KG, Mills DA, Medzhitov RM. The human gut microbiota and undernutrition. Sci Transl Med. 2012 Jun 6;4(137):137ps12. doi: 10.1126/scitranslmed.3004347. PMID 22674549
- [Background] Garrido D, Ruiz-Moyano S, Mills DA. Release and utilization of N-acetyl-D-glucosamine from human milk oligosaccharides by Bifidobacterium longum subsp. infantis. Anaerobe. 2012 Aug;18(4):430-5. doi: 10.1016/j.anaerobe.2012.04.012. Epub 2012 May 9. PMID 22579845
- [Background] Chichlowski M, De Lartigue G, German JB, Raybould HE, Mills DA. Bifidobacteria isolated from infants and cultured on human milk oligosaccharides affect intestinal epithelial function. J Pediatr Gastroenterol Nutr. 2012 Sep;55(3):321-7. doi: 10.1097/MPG.0b013e31824fb899. PMID 22383026
- [Background] Garrido D, Kim JH, German JB, Raybould HE, Mills DA. Oligosaccharide binding proteins from Bifidobacterium longum subsp. infantis reveal a preference for host glycans. PLoS One. 2011 Mar 15;6(3):e17315. doi: 10.1371/journal.pone.0017315. PMID 21423604
- [Background] Barboza M, Sela DA, Pirim C, Locascio RG, Freeman SL, German JB, Mills DA, Lebrilla CB. Glycoprofiling bifidobacterial consumption of galacto-oligosaccharides by mass spectrometry reveals strain-specific, preferential consumption of glycans. Appl Environ Microbiol. 2009 Dec;75(23):7319-25. doi: 10.1128/AEM.00842-09. Epub 2009 Oct 2. PMID 19801485
- [Result] Barboza M, Pinzon J, Wickramasinghe S, Froehlich JW, Moeller I, Smilowitz JT, Ruhaak LR, Huang J, Lonnerdal B, German JB, Medrano JF, Weimer BC, Lebrilla CB. Glycosylation of human milk lactoferrin exhibits dynamic changes during early lactation enhancing its role in pathogenic bacteria-host interactions. Mol Cell Proteomics. 2012 Jun;11(6):M111.015248. doi: 10.1074/mcp.M111.015248. Epub 2012 Jan 19. PMID 22261723
- [Result] Argov-Argaman N, Smilowitz JT, Bricarello DA, Barboza M, Lerno L, Froehlich JW, Lee H, Zivkovic AM, Lemay DG, Freeman S, Lebrilla CB, Parikh AN, German JB. Lactosomes: structural and compositional classification of unique nanometer-sized protein lipid particles of human milk. J Agric Food Chem. 2010 Nov 10;58(21):11234-42. doi: 10.1021/jf102495s. Epub 2010 Oct 6. PMID 20925428
- [Result] Yang Y, Rader E, Peters-Carr M, Bent RC, Smilowitz JT, Guillemin K, Rader B. Ontogeny of alkaline phosphatase activity in infant intestines and breast milk. BMC Pediatr. 2019 Jan 3;19(1):2. doi: 10.1186/s12887-018-1379-1. PMID 30606146
- [Result] Nijman RM, Liu Y, Bunyatratchata A, Smilowitz JT, Stahl B, Barile D. Characterization and Quantification of Oligosaccharides in Human Milk and Infant Formula. J Agric Food Chem. 2018 Jul 5;66(26):6851-6859. doi: 10.1021/acs.jafc.8b01515. Epub 2018 Jun 20. PMID 29799744
- [Result] Bever CS, Rand AA, Nording M, Taft D, Kalanetra KM, Mills DA, Breck MA, Smilowitz JT, German JB, Hammock BD. Effects of triclosan in breast milk on the infant fecal microbiome. Chemosphere. 2018 Jul;203:467-473. doi: 10.1016/j.chemosphere.2018.03.186. Epub 2018 Mar 28. PMID 29635158
- [Result] Xu G, Davis JC, Goonatilleke E, Smilowitz JT, German JB, Lebrilla CB. Absolute Quantitation of Human Milk Oligosaccharides Reveals Phenotypic Variations during Lactation. J Nutr. 2017 Jan;147(1):117-124. doi: 10.3945/jn.116.238279. Epub 2016 Oct 19. PMID 27798342
- [Result] Huang J, Kailemia MJ, Goonatilleke E, Parker EA, Hong Q, Sabia R, Smilowitz JT, German JB, Lebrilla CB. Quantitation of human milk proteins and their glycoforms using multiple reaction monitoring (MRM). Anal Bioanal Chem. 2017 Jan;409(2):589-606. doi: 10.1007/s00216-016-0029-4. Epub 2016 Oct 29. PMID 27796459
- [Result] Davis JC, Totten SM, Huang JO, Nagshbandi S, Kirmiz N, Garrido DA, Lewis ZT, Wu LD, Smilowitz JT, German JB, Mills DA, Lebrilla CB. Identification of Oligosaccharides in Feces of Breast-fed Infants and Their Correlation with the Gut Microbial Community. Mol Cell Proteomics. 2016 Sep;15(9):2987-3002. doi: 10.1074/mcp.M116.060665. Epub 2016 Jul 19. PMID 27435585
- [Result] Napoli E, Ross-Inta C, Song G, Wong S, Hagerman R, Gane LW, Smilowitz JT, Tassone F, Giulivi C. Premutation in the Fragile X Mental Retardation 1 (FMR1) Gene Affects Maternal Zn-milk and Perinatal Brain Bioenergetics and Scaffolding. Front Neurosci. 2016 Apr 19;10:159. doi: 10.3389/fnins.2016.00159. eCollection 2016. PMID 27147951
- [Result] Lewis ZT, Davis JC, Smilowitz JT, German JB, Lebrilla CB, Mills DA. The impact of freeze-drying infant fecal samples on measures of their bacterial community profiles and milk-derived oligosaccharide content. PeerJ. 2016 Jan 21;4:e1612. doi: 10.7717/peerj.1612. eCollection 2016. PMID 26819854
- [Result] Goldsmith F, O'Sullivan A, Smilowitz JT, Freeman SL. Lactation and Intestinal Microbiota: How Early Diet Shapes the Infant Gut. J Mammary Gland Biol Neoplasia. 2015 Dec;20(3-4):149-58. doi: 10.1007/s10911-015-9335-2. Epub 2015 Jul 31. PMID 26227402
- [Result] Spevacek AR, Smilowitz JT, Chin EL, Underwood MA, German JB, Slupsky CM. Infant Maturity at Birth Reveals Minor Differences in the Maternal Milk Metabolome in the First Month of Lactation. J Nutr. 2015 Aug;145(8):1698-708. doi: 10.3945/jn.115.210252. Epub 2015 Jun 3. PMID 26041675
- [Result] Beck KL, Weber D, Phinney BS, Smilowitz JT, Hinde K, Lonnerdal B, Korf I, Lemay DG. Comparative Proteomics of Human and Macaque Milk Reveals Species-Specific Nutrition during Postnatal Development. J Proteome Res. 2015 May 1;14(5):2143-57. doi: 10.1021/pr501243m. Epub 2015 Apr 6. PMID 25757574
- [Result] Huang J, Guerrero A, Parker E, Strum JS, Smilowitz JT, German JB, Lebrilla CB. Site-specific glycosylation of secretory immunoglobulin A from human colostrum. J Proteome Res. 2015 Mar 6;14(3):1335-49. doi: 10.1021/pr500826q. Epub 2015 Feb 11. PMID 25629924
- [Result] Dallas DC, Smink CJ, Robinson RC, Tian T, Guerrero A, Parker EA, Smilowitz JT, Hettinga KA, Underwood MA, Lebrilla CB, German JB, Barile D. Endogenous human milk peptide release is greater after preterm birth than term birth. J Nutr. 2015 Mar;145(3):425-33. doi: 10.3945/jn.114.203646. Epub 2014 Dec 24. PMID 25540406
- [Result] Grapov D, Lemay DG, Weber D, Phinney BS, Azulay Chertok IR, Gho DS, German JB, Smilowitz JT. The human colostrum whey proteome is altered in gestational diabetes mellitus. J Proteome Res. 2015 Jan 2;14(1):512-20. doi: 10.1021/pr500818d. Epub 2014 Dec 1. PMID 25338220
- [Result] Lewis ZT, Totten SM, Smilowitz JT, Popovic M, Parker E, Lemay DG, Van Tassell ML, Miller MJ, Jin YS, German JB, Lebrilla CB, Mills DA. Maternal fucosyltransferase 2 status affects the gut bifidobacterial communities of breastfed infants. Microbiome. 2015 Apr 10;3:13. doi: 10.1186/s40168-015-0071-z. eCollection 2015. PMID 25922665
- [Result] O'Sullivan A, Farver M, Smilowitz JT. The Influence of Early Infant-Feeding Practices on the Intestinal Microbiome and Body Composition in Infants. Nutr Metab Insights. 2015 Dec 16;8(Suppl 1):1-9. doi: 10.4137/NMI.S29530. eCollection 2015. PMID 26715853
- [Result] Totten SM, Wu LD, Parker EA, Davis JC, Hua S, Stroble C, Ruhaak LR, Smilowitz JT, German JB, Lebrilla CB. Rapid-throughput glycomics applied to human milk oligosaccharide profiling for large human studies. Anal Bioanal Chem. 2014 Dec;406(30):7925-35. doi: 10.1007/s00216-014-8261-2. Epub 2014 Oct 31. PMID 25358913
- [Result] Khaldi N, Vijayakumar V, Dallas DC, Guerrero A, Wickramasinghe S, Smilowitz JT, Medrano JF, Lebrilla CB, Shields DC, German JB. Predicting the important enzymes in human breast milk digestion. J Agric Food Chem. 2014 Jul 23;62(29):7225-32. doi: 10.1021/jf405601e. Epub 2014 Jul 10. PMID 24620897
- [Result] Smilowitz JT, Gho DS, Mirmiran M, German JB, Underwood MA. Rapid measurement of human milk macronutrients in the neonatal intensive care unit: accuracy and precision of fourier transform mid-infrared spectroscopy. J Hum Lact. 2014 May;30(2):180-9. doi: 10.1177/0890334413517941. Epub 2014 Jan 14. PMID 24423984
- [Result] Hong Q, Ruhaak LR, Totten SM, Smilowitz JT, German JB, Lebrilla CB. Label-free absolute quantitation of oligosaccharides using multiple reaction monitoring. Anal Chem. 2014 Mar 4;86(5):2640-7. doi: 10.1021/ac404006z. Epub 2014 Feb 20. PMID 24502421
- [Result] Huang J, Lee H, Zivkovic AM, Smilowitz JT, Rivera N, German JB, Lebrilla CB. Glycomic analysis of high density lipoprotein shows a highly sialylated particle. J Proteome Res. 2014 Feb 7;13(2):681-91. doi: 10.1021/pr4012393. Epub 2014 Jan 21. PMID 24417605
- [Result] Smilowitz JT, Lebrilla CB, Mills DA, German JB, Freeman SL. Breast milk oligosaccharides: structure-function relationships in the neonate. Annu Rev Nutr. 2014;34:143-69. doi: 10.1146/annurev-nutr-071813-105721. Epub 2014 May 15. PMID 24850388
- [Result] Lemay DG, Hovey RC, Hartono SR, Hinde K, Smilowitz JT, Ventimiglia F, Schmidt KA, Lee JW, Islas-Trejo A, Silva PI, Korf I, Medrano JF, Barry PA, German JB. Sequencing the transcriptome of milk production: milk trumps mammary tissue. BMC Genomics. 2013 Dec 12;14:872. doi: 10.1186/1471-2164-14-872. PMID 24330573
- [Result] Smilowitz JT, Totten SM, Huang J, Grapov D, Durham HA, Lammi-Keefe CJ, Lebrilla C, German JB. Human milk secretory immunoglobulin a and lactoferrin N-glycans are altered in women with gestational diabetes mellitus. J Nutr. 2013 Dec;143(12):1906-12. doi: 10.3945/jn.113.180695. Epub 2013 Sep 18. PMID 24047700
- [Result] Smilowitz JT, O'Sullivan A, Barile D, German JB, Lonnerdal B, Slupsky CM. The human milk metabolome reveals diverse oligosaccharide profiles. J Nutr. 2013 Nov;143(11):1709-18. doi: 10.3945/jn.113.178772. Epub 2013 Sep 11. PMID 24027187
- [Result] Ruiz-Moyano S, Totten SM, Garrido DA, Smilowitz JT, German JB, Lebrilla CB, Mills DA. Variation in consumption of human milk oligosaccharides by infant gut-associated strains of Bifidobacterium breve. Appl Environ Microbiol. 2013 Oct;79(19):6040-9. doi: 10.1128/AEM.01843-13. Epub 2013 Jul 26. PMID 23892749
- [Result] Dallas DC, Guerrero A, Khaldi N, Castillo PA, Martin WF, Smilowitz JT, Bevins CL, Barile D, German JB, Lebrilla CB. Extensive in vivo human milk peptidomics reveals specific proteolysis yielding protective antimicrobial peptides. J Proteome Res. 2013 May 3;12(5):2295-304. doi: 10.1021/pr400212z. Epub 2013 Apr 24. PMID 23586814
- [Result] Dallas DC, Martin WF, Strum JS, Zivkovic AM, Smilowitz JT, Underwood MA, Affolter M, Lebrilla CB, German JB. N-linked glycan profiling of mature human milk by high-performance microfluidic chip liquid chromatography time-of-flight tandem mass spectrometry. J Agric Food Chem. 2011 Apr 27;59(8):4255-63. doi: 10.1021/jf104681p. Epub 2011 Mar 18. PMID 21384928
- [Derived] Goonatilleke E, Huang J, Xu G, Wu L, Smilowitz JT, German JB, Lebrilla CB. Human Milk Proteins and Their Glycosylation Exhibit Quantitative Dynamic Variations during Lactation. J Nutr. 2019 Aug 1;149(8):1317-1325. doi: 10.1093/jn/nxz086. PMID 31098625
- See also: Details for this research project is available through the UC Davis Foods for Health Institute website — https://ffhi.ucdavis.edu/human-studies